CLINICAL TRIAL: NCT02498093
Title: Maximal Strength Training in Patients Undergoing Total Hip Arthroplasty: Implementing Evidence Based Rehabilitation Into Clinical Practice, and the Influence of Supervised Training
Brief Title: Maximal Strength Training in Patients Undergoing Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2010/3373
Record Dates: First submitted 2015-07-08; First posted 2015-07-15 (Estimated); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Muscle Weakness
Keywords: Resistance training; Arthroplasty, Replacement, Hip; Professional-Patient Relations; Evidence-based practice
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maximal strength training (Experimental): Maximal strength training supervised by a physiotherapist
  Interventions: Behavioral: Maximal strength training
- Control (Active Comparator): Conventional rehabilitation supervised by a physiotherapist
  Interventions: Behavioral: conventional rehabilitation

INTERVENTIONS:
Behavioral: Maximal strength training
  Arms: Maximal strength training
Behavioral: conventional rehabilitation
  Arms: Control

SUMMARY:
Conventional rehabilitation after total hip arthroplasty (THA) does not seem to restore muscular strength or walking speed. Three-5 years after surgery patients are still not fully rehabilitated. This study evaluates the effects of maximal strength training on the muscular strength in leg press and abduction in patients undergoing THA. Aim of the study is to increase the patients physical function through evidence-based rehabilitation in clinical practice, with gradually less supervision.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for total hip arthroplasty (THA)
* living nearby Trondheim
* diagnosis of primary osteoarthritis as the main cause for elective THA
* ASA score of I-III (stable)

Exclusion Criteria:

* muscular or skeletal disease which might influence the training and/or physical testing performance
* communication difficulties
* postoperatively discharged to a rehabilitation institution
* THA in the bilateral hip that is not fully rehabilitated.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Muscular strength | 3 months
  leg press (kg), abduction (kg)
Muscular strength | 6 months
  leg press (kg), abduction (kg)
muscular strength | 1 year
  leg press (kg), abduction (kg)

SECONDARY OUTCOMES:
Physical function | up to 1 year
  Harris hip score, 6 min walking test
Bone mineral density | up to 1 year
  Dual X-ray absorptiometry (DXA)

CONTACTS AND LOCATIONS:
Overall Officials: Lars Jacob Stovner, prof, Study Director — Norwegian University of Science and Technology
Locations (1):
- Department of Neuroscience, Faculty of Medicine, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Winther SB, Foss OA, Klaksvik J, Husby VS. Pain and load progression following an early maximal strength training program in total hip- and knee arthroplasty patients. J Orthop Surg (Hong Kong). 2020 Jan-Apr;28(2):2309499020916392. doi: 10.1177/2309499020916392. PMID 32301372
- [Result] Winther SB, Foss OA, Husby OS, Wik TS, Klaksvik J, Husby VS. A randomized controlled trial on maximal strength training in 60 patients undergoing total hip arthroplasty. Acta Orthop. 2018 Jun;89(3):295-301. doi: 10.1080/17453674.2018.1441362. Epub 2018 Mar 1. PMID 29493347